CLINICAL TRIAL: NCT01235676
Title: Is it Possible to Reduce the Number of Macrosomic Infants With Abundant Fat Tissue by Lifestyle Intervention During Pregnancy ?
Brief Title: Tissue Composition of Newborn Infants of Obese and Lean Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ole Pryds, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DEXA-2650
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Obesity
Keywords: obesity; lifestyle; pregnancy; newborn infant
MeSH Terms: conditions — Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet (Experimental): Calorie restriction to reduce weight gain
  Interventions: Behavioral: diet
- Exercise (Experimental): Exercise to reduce weight gain
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: diet — calorie restriction to reduce weight gain
  Arms: Diet
Behavioral: Exercise — Exercise to reduce weight gain
  Arms: Exercise

SUMMARY:
0-hypothesis: the tissue composition of newborn infants is not modified by lifestyle intervention during pregnancy

DETAILED DESCRIPTION:
Obese pregnant women (BMI > 30) are randomized to exercise, diet or control (1:1:1) in order to reduce weight gain during pregnancy. Shortly after birth, tissue composition will be measured (DEXA)in 200 infants (65 from each group). The amount of fat tissue is subsequently analyzed between the groups and compared to results from another 65 infants of lean mothers

ELIGIBILITY:
Inclusion Criteria:

Healthy term neonates Informed and written consent from both parents -

Exclusion Criteria:

Sick or preterm infants No consent

-

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 270 (Actual)
Dates: Start 2010-02; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
amount of fat tissue | at birth

SECONDARY OUTCOMES:
birth weight | at birth

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark